CLINICAL TRIAL: NCT06042153
Title: Semaglutide for Dialysis-Treated Patients - a Glucose Time in Range Study- DIALYSIS-TIR Study
Brief Title: DIALYSIS-TIR Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Ildiko Lingvay, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2022-0786
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; End Stage Renal Disease on Dialysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double-blind, parallel-group, placebo-controlled, trial comparing semaglutide subcutaneously weekly versus matched placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization and each dispensation will be performed by blinded study staff using an electronic system coded with the randomization code, to ensure all study personnel remains blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Semaglutide (Experimental): Participants will receive semaglutide as an adjunct to standard-of-care.
  Interventions: Drug: Semaglutide
- Arm 2- Placebo (Placebo Comparator): Participants will receive placebo (semaglutide) as an adjunct to standard-of-care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide will be injected into a skin fold, in the stomach, thigh or upper arm once a week at the same day of the week (to the extent possible) throughout the trial. Subjects will start semaglutide treatment at 0.25 mg; dose will gradually be increased every 4 weeks up to 1.0 mg.
  Arms: Arm 1 - Semaglutide
Drug: Placebo — Placebo will be injected into a skin fold, in the stomach, thigh or upper arm once a week at the same day of the week (to the extent possible) throughout the trial. Participants will receive placebo at an equivalent dose to semaglutide.
  Arms: Arm 2- Placebo

SUMMARY:
This study will look at control of blood sugar levels in persons with type 2 diabetes mellitus currently on chronic dialysis. Researchers will compare blood sugar levels in people taking semaglutide to people taking "dummy" medicine. The treatment participants get will be decided randomly.

Participants will need to inject the study medication once a week. The study will last for 1 year and a month. Participants will be asked to wear a sensor that measures blood sugar levels for a period of 10 days at five different time points during the study.

DETAILED DESCRIPTION:
The researchers also have a Data Safety Monitoring Plan in place.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent before any trial-related activities. Trial-related activities are any procedures that are carried out as a part of trial, including activities to determine suitability for the trial.
2. Male or female Adults (age > 18 years at the time of signing the consent)
3. Type 2 diabetes mellitus diagnosed > 6 months prior to screening
4. On current chronic treatment with Hemodialysis or Peritoneal dialysis for > 6 months prior to screening
5. Current treatment with any glucose lowering pharmacotherapy, at a stable dose for at least 30 days. DPP-4 Inhibitors will be allowed at study entry and will be stopped at randomization.
6. Minimum of 80% valid data on the 10-day Continuous Glucose Monitor download
7. Time in Range 15 to 60%

Exclusion Criteria:

1. BMI < 23 kg/m2 at screening
2. Current (within the past 90 days of screening) use of any GLP-1 RA
3. Personal or family history of medullary thyroid cancer or Multiple Endocrine Neoplasia type 2
4. Known or suspected hypersensitivity to GLP-1 RA (trial medication(s), excipients, or related products)
5. Pregnant, breast-feeding or the intention of becoming pregnant, or not using effective contraceptive measures
6. Active weight loss, defined as weight loss of >5% of body weight in the past 3 months
7. Current participation in other interventional trials or last dose of any investigational product within 4 half- lives at the time of randomization
8. Any medical condition which in the judgement of the investigator precludes safe participation in the trial (includes, but not limited to active neoplasm, severe heart failure, recent cardiovascular event, severe frailty, planned cardiac or vascular surgeries on the day of screening etc)
9. If weight loss is not desired by the participant, or if the provider or investigator considers intentional weight loss to be detrimental to the health of the participant
10. Other or secondary forms of diabetes (like type 1 diabetes, pancreatogenic diabetes mellitus, MODY, LADA, drug induced, etc.)
11. Current diagnosis of gastroparesis or enteropathywhich in the opinion of investigator precludes safe treatment with GLP-1 RA.
12. Hypoglycaemia unawareness, or history of frequent or severe hypoglycaemia (in the opinion of the investigator)
13. Personal history of chronic pancreatitis, or acute pancreatitis within 180 days of screening
14. Known current uncontrolled or unstable retinopathy (by medical history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in TIR (70-180 mg/dl) | Baseline, 52 weeks
  Measured in percentage by Continuous glucose monitor (CGM)

SECONDARY OUTCOMES:
Change in Time in high range (180-250 mg/dl) | Baseline, 52 weeks
  Measured in percentage by Continuous glucose monitor (CGM)
Change in Time in very high range (>250 mg/dl) | Baseline, 52 weeks
  Measured in percentage by Continuous glucose monitor (CGM)
Change in Time in low range (54-69 mg/dl) | Baseline, 52 weeks
  Measured in percentage by Continuous glucose monitor (CGM)
Change in Time in very low range (<54 mg/dl) | Baseline, 52 weeks
  Measured in percentage by Continuous glucose monitor (CGM)
Proportion of participants with TIR 70-180 mg/dl for 70% of the day | 52 weeks
  Measured in percentage by CGM
Proportion of participants with TIR 70-180 mg/dl with more than equal to 5% improvement from baseline | 52 weeks
  Measured in percentage by CGM
Proportion of participants with Time below range <70 mg/dL for <4% of each day | 52 weeks
  Measured in percentage by CGM
Proportion of participants with Time below range <54 mg/dL for <1% of each day | 52 weeks
  Measured in percentage by CGM
Proportion of participants with Time above range >180 mg/dL for <25% of each day | 52 weeks
  Measured in percentage by CGM
Change in haemoglobin A1c (HbA1c) | Baseline, 52 weeks
  Measured in percentage
Total daily dose of insulin | 52 weeks
  Measured as units/day
Number of oral glucose lowering agents | 52 weeks
  Measured as count
Proportion of participants with >10 points improvement in % TIR 70-180 mg/dL without an increase in time below range <54 mg/dL of >0.5% | 52 weeks
  Measured in percentage
Proportion of participants with mean glucose <154 mg/dL and <1% time below range <54 mg/dL | 52 weeks
  Measured in percentage
Number of participants with Severe hypoglycemia | 52 weeks
  Measured in count
Change in body weight | Baseline, 52 weeks
  Measured in kilograms
Change in waist circumference | Baseline, 52 weeks
  Measured in centimeters
Change in percentage total body fat | Baseline, 52 weeks
  Measured in percentage
Change in percentage lean mass | Baseline, 52 weeks
  Measured in percentage
Change in Inter-dialysis weight gain | Baseline, 52 weeks
  Measured in kilograms
Number of participants hospitalized | 52 weeks
  Measured in count
Total number of days spent in hospital | 52 weeks
  Measured in count
Total score of Diabetes Treatment Satisfaction questionnaire | 52 weeks
  Patient reported outcomes is assessed by Diabetes Treatment Satisfaction Score questionnaire which assesses patient satisfaction with diabetes treatment. It is composed of eight questions, each of which is scored by patients on a scale ranging from zero (e.g., "very dissatisfied", "very inconvenient") to six (e.g., "very satisfied", "very convenient"). Treatment satisfaction is assessed as the sum of the scores of the six questions on the first factor, with a higher score indicating higher treatment satisfaction.
Total score of EQ-5D-5L | 52 weeks
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. Possible scores range from 0-100, where higher score indicate better outcome
Total score of Kidney disease QoL short form | 52 weeks
  The KDQOL-SF is a self-report measure developed for individuals with kidney disease and those on dialysis. It is a shorter version of a measure developed by the same authors. It includes 43 kidney disease-targeted items, such as the effects of the disease of activities of daily living, work status, and social interaction, and 36 items that provide a measure of physical and mental health, and 1 overall health rating item ranging from 0 ("worst possible health") to 10 ("best possible health.").

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Lingvay, MD, MPH, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (5):
- United States (5):
  - University of North Carolina, Chapel Hill, North Carolina
  - Davita UT Southwestern - Oak Cliff, Dallas, Texas
  - DaVita UT Southwestern - East Dallas, Dallas, Texas
  - DaVita UT Southwestern - Preston, Dallas, Texas
  - DaVita UT Southwestern - Irving, Irving, Texas

IPD SHARING:
Plan to Share IPD: No